CLINICAL TRIAL: NCT02702999
Title: Determination of Abnormal Fetal Growth or Amniotic Fluid With Third Trimester Ultrasounds in Uncomplicated Pregnancies: A Randomized Trial (UP Trial)
Brief Title: Determination of Abnormal Fetal Growth or Amniotic Fluid With Third Trimester Ultrasounds in Uncomplicated Pregnancies: A Randomized Trial
Acronym: UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Olaide Ashimi Balogun, Fellow, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-16-0084
Record Dates: First submitted 2016-02-25; First posted 2016-03-09 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Uncomplicated Pregnancy; Abnormal Fetal Growth or Fluid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine third trimester care (Active Comparator): Routine third trimester care with clinically-indicated ultrasound (control)
  Interventions: Device: Clinically-indicated ultrasound
- Serial third trimester ultrasound (Experimental): Ultrasound evaluation for fetal growth and amniotic fluid will be performed every 4 weeks starting at 30 weeks (intervention group). Thus, if they continue to term, there will be 3 additional ultrasounds exams (30, 34 and 38 weeks).
  Interventions: Device: Serial third trimester ultrasound

INTERVENTIONS:
Device: Clinically-indicated ultrasound — Routine third trimester care with clinically-indicated ultrasound (control)
  Arms: Routine third trimester care
Device: Serial third trimester ultrasound — Ultrasound evaluation for fetal growth and amniotic fluid will be performed every 4 weeks starting at 30 weeks (intervention group). Thus, if they continue to term, there will be 3 additional ultrasounds exams (30, 34 and 38 weeks).
  Arms: Serial third trimester ultrasound

SUMMARY:
The purpose of this study is to see whether women at a gestational age of 30 weeks or more without comorbidities, does performance of serial 3rd trimester growth ultrasounds increase the frequency of identifying abnormalities in fetal growth or amniotic fluid, when compared with women who only receive indicated ultrasounds?

ELIGIBILITY:
Inclusion Criteria:

* Maternal age of 18 at the time of consent
* Singleton gestation

Exclusion Criteria:

* First sonographic examination after 20 weeks
* Women with any of the following co-morbidities: Autoimmune disorders (antiphospholipid antibody, lupus, rheumatoid arthritis, scleroderma), Cerclage in the index pregnancy, Diabetes mellitus-gestational or pre-gestational, Hematologic disorders (coagulation defects, sickle cell disease, thrombocytopenia, thrombophilia), Hypertension (chronic or pregnancy induced) before enrollment, HIV (human immunodeficiency virus), Institutionalized individuals (prisoners), Prior obstetric history of: [1) intrauterine growth restriction, 2) preterm birth before 34 weeks, 3) severe preeclampsia], eclampsia, HELLP syndrome, and 4) stillbirth after 24 weeks or neonatal death, Preterm labor or ruptured membranes before enrollment, Psychiatric disorder (bipolar, depression) on medication, Placenta previa / 3rd trimester bleeding, Renal insufficiency (serum creatinine > 1.5 mg/dL), Restrictive lung disease, Fetal red blood cell isoimmunization, Seizure disorder on medication, Thyroid disease on medication, Body Mass Index (BMI) above 40 kg/m2
* Major fetal Anomaly including: anencephaly, spina bifida, bilateral renal agenesis, cystic hygroma with hydrops, diaphragmatic hernia, or congenital heart defects
* Unable to understand consent in English or Spanish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2016-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olaide A Ashimi Balogun, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - UT Physicians, Bellaire, Texas
  - University of Texas at Houston Health Science Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ashimi Balogun O, Sibai BM, Pedroza C, Blackwell SC, Barrett TL, Chauhan SP. Serial Third-Trimester Ultrasonography Compared With Routine Care in Uncomplicated Pregnancies: A Randomized Controlled Trial. Obstet Gynecol. 2018 Dec;132(6):1358-1367. doi: 10.1097/AOG.0000000000002970. PMID 30399092

RESULTS

PARTICIPANT FLOW:
Groups:
- Serial Third Trimester Ultrasound: Serial third trimester ultrasound: Ultrasound evaluation for fetal growth and amniotic fluid will be performed every 4 weeks starting at 30 weeks. Thus, if they continue to term, there will be 3 additional ultrasounds exams (30, 34 and 38 weeks).
Period: Overall Study
Arm/Group | Routine Third Trimester Care | Serial Third Trimester Ultrasound
Started | 102 | 104
Completed | 102 | 104
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Third Trimester Care | Serial Third Trimester Ultrasound | Total
Number analyzed (Participants) | 102 | 104 | 206
Age, Customized [Count of Participants; unit: Participants]
  less than 20 years old | 5 | 10 | 15
  20 to 34 years old | 87 | 82 | 169
  greater than or equal to 35 years old | 10 | 12 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 104 | 206
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black | 32 | 34 | 66
  Race/Ethnicity: White | 23 | 25 | 48
  Race/Ethnicity: Hispanic | 20 | 22 | 42
  Race/Ethnicity: Other | 27 | 23 | 50
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 102 | 104 | 206
Nulliparity (never given birth) [Count of Participants; unit: Participants] | 43 | 39 | 82
Insurance [Count of Participants; unit: Participants]
  Medicaid | 66 | 69 | 135
  Private Insurance | 36 | 35 | 71
Body Mass Index (BMI) at first prenatal visit [Count of Participants; unit: Participants]
  less than 30 kg/m^2 | 74 | 77 | 151
  30 to 39.9 kg/m^2 | 28 | 27 | 55
Time of first ultrasound exam [Mean (Standard Deviation); unit: weeks] | 12.9 (4.3) | 12.9 (4.3) | 12.9 (4.3)
Gestational Age at Randomization [Mean (Standard Deviation); unit: weeks] | 29.2 (1.0) | 29.0 (1.1) | 29.1 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Fetal Growth Restriction
Time Frame: 30 to 38 weeks gestational age
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Third Trimester Care | Serial Third Trimester Ultrasound
Number analyzed (Participants) | 102 | 104
Participants | 2 | 8
Statistical Analysis 1: Comparison: Routine Third Trimester Care vs Serial Third Trimester Ultrasound; Test type: Superiority; Risk Ratio (RR) = 3.9, 95% CI 2-sided [0.9 to 18.0] — The intervention arm and control arm were compared using a log binomial (or Poisson in case of nonconvergence) model with the intervention arm as a covariate to estimate relative risk and 95% confidence interval (CI)

2. Primary Outcome: Number of Participants With Large for Gestational Age Fetuses
Time Frame: 30 to 38 weeks gestational age
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Third Trimester Care | Serial Third Trimester Ultrasound
Number analyzed (Participants) | 102 | 104
Participants | 2 | 8
Statistical Analysis 1: Comparison: Routine Third Trimester Care vs Serial Third Trimester Ultrasound; Test type: Superiority; Risk Ratio (RR) = 3.9, 95% CI 2-sided [0.9 to 18.0] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Number of Participates With Oligohydraminos
Description: Oligohydramnios is a condition in pregnancy characterized by a deficiency of amniotic fluid. Amniotic fluid was assessed using the amniotic fluid index (AFI) or maximum vertical pocket (MVP). Oligohydramnios was defined as AFI less than or equal to 5.0 cm or MVP less than or equal to 2.0 cm.
  AFI is the sum of the vertical length of the deepest, unobstructed pocket of amniotic fluid in each of the 4 quadrants of the pregnant uterus. An AFI of less than or equal to 5cm is considered low amniotic fluid, and an AFI greater than or equal to 24cm is considered high amniotic fluid.
  MVP is the vertical length of the single deepest pocket of amniotic fluid. An MVP less than or equal to 2cm is considered to be low amniotic fluid and an MVP of 8cm or greater is considered to be high amniotic fluid.
  Both low and high amniotic fluid levels are worse outcomes than having normal amniotic fluid levels.
Time Frame: 30 to 38 weeks gestational age
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Third Trimester Care | Serial Third Trimester Ultrasound
Number analyzed (Participants) | 102 | 104
Participants | 2 | 4
Statistical Analysis 1: Comparison: Routine Third Trimester Care vs Serial Third Trimester Ultrasound; Test type: Superiority; Risk Ratio (RR) = 1.9, 95% CI 2-sided [0.4 to 10.5] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Number of Participates With Polyhydraminos
Description: Polyhydraminos is a condition in pregnancy characterized by an excess of amniotic fluid. Amniotic fluid was assessed using either the amniotic fluid index (AFI) or maximum vertical pocket (MVP). Polyhydramnios was defined as AFI greater than or equal to 24.0 cm or MVP greater than or equal to 8.0 cm.
  AFI is the sum of the vertical length of the deepest, unobstructed pocket of amniotic fluid in each of the 4 quadrants of the pregnant uterus. An AFI of less than or equal to 5cm is considered low amniotic fluid, and an AFI greater than or equal to 24cm is considered high amniotic fluid.
  MVP is the vertical length of the single deepest pocket of amniotic fluid. An MVP less than or equal to 2cm is considered to be low amniotic fluid and an MVP of 8cm or greater is considered to be high amniotic fluid.
  Both low and high amniotic fluid levels are worse outcomes than having normal amniotic fluid levels.
Time Frame: 30 to 38 weeks gestational age
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Third Trimester Care | Serial Third Trimester Ultrasound
Number analyzed (Participants) | 102 | 104
Participants | 2 | 11
Statistical Analysis 1: Comparison: Routine Third Trimester Care vs Serial Third Trimester Ultrasound; Test type: Superiority; Risk Ratio (RR) = 5.4, 95% CI 2-sided [1.2 to 23.7] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants With Composite Neonatal Morbidity
Description: Composite Neonatal Morbidity is defined as the presence of one or more of the following: 1) Apgar score < 5 at 5 min; 2) umbilical arterial pH < 7.00; 3) intraventricular hemorrhage grade III or IV; 4) periventricular leukomalacia; 5) intubation for over 24 hrs; 6) necrotizing enterocolitis grade 2 or 3; 7) stillbirth; or 8) death within 28 days of birth.
Time Frame: From time of delivery to 28 days after delivery
Population: One patient in the routine third trimester care group delivered in an outside hospital, and the data was not available.
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Third Trimester Care | Serial Third Trimester Ultrasound
Number analyzed (Participants) | 101 | 104
Participants | 4 | 1
Statistical Analysis 1: Comparison: Routine Third Trimester Care vs Serial Third Trimester Ultrasound; Test type: Superiority; Risk Ratio (RR) = 0.2, 95% CI 2-sided [0.03 to 2.1] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Participants With Composite Maternal Morbidity
Description: Composite Maternal Morbidity is defined as the presence of one of more of the following: 1) chorioamnionitis; 2) cesarean delivery in labor; 3) wound infection; 4) transfusion; 5) deep venous thrombus or pulmonary embolism; 6) admission to intensive care unit; 7) postpartum hemorrhage; or 8) death.
Time Frame: From time of delivery to discharge (average time of discharge is 4 days after delivery)
Population: One patient in the routine third trimester care group delivered in an outside hospital, and the data was not available.
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Third Trimester Care | Serial Third Trimester Ultrasound
Number analyzed (Participants) | 101 | 104
Participants | 9 | 9
Statistical Analysis 1: Comparison: Routine Third Trimester Care vs Serial Third Trimester Ultrasound; Test type: Superiority; Risk Ratio (RR) = 1.0, 95% CI 2-sided [0.4 to 2.3] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From time of delivery to discharge (average time of discharge is 4 days after delivery)
Description: None of the below-reported adverse events were deemed to be related to the study interventions.
Arm/Group | Routine Third Trimester Care | Serial Third Trimester Ultrasound
All-Cause Mortality (participants affected / at risk) | 1/102 | 0/104
Serious Adverse Events (participants affected / at risk) | 1/102 | 0/104
Other Adverse Events (participants affected / at risk) | 25/102 | 22/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Routine Third Trimester Care (N=102) | Serial Third Trimester Ultrasound (N=104)
Neonatal death (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Routine Third Trimester Care (N=102) | Serial Third Trimester Ultrasound (N=104)
gestational hypertension (GHTN)/preeclampsia (Pregnancy, puerperium and perinatal conditions) | 15 (15) | 21 (21)
Decreased fetal movement (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 3 (3)
Preterm labor (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 3 (3)
Premature rupture of membranes (PROM) (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3)
Cholestasis, pyelonephritis, fall, or fetal ventricular tachycardia (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 2 (2)
Chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 5 (5)
Cesarean delivery in labor (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 5 (5)
Postpartum Hemorrhage (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2)
Transfusion (maternal) (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1)
Wound infection (maternal) (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Apgar score < 5 at 5 min (General disorders) | 1 (1) | 0 (0)
Umbilical arterial pH < 7.00 (General disorders) | 2 (2) | 0 (0)
Intubation over 24 hours (infant) (General disorders) | 1 (1) | 1 (1)
Intraventricular hemorrhage (IVH) grade III or IV (infant) (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
not powered to detect differences in neonatal outcomes; all sonographic exams were done by a Registered Diagnostic Medical Sonographer (RDMS), and thus findings may not apply to those with sonographic exams done by clinician

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT02702999/Prot_SAP_000.pdf